CLINICAL TRIAL: NCT03157349
Title: Immediate and Short-term Effect of Biofreeze® Versus Placebo on Acute Neck Pain, Disability, and Range of Motion
Brief Title: Effect of Biofreeze® Versus Placebo on Acute Neck Pain, Disability, and Range of Motion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sport and Spine Rehab Clinical Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Neck BFvP
Record Dates: First submitted 2017-05-12; First posted 2017-05-17 (Actual); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Acute Pain; Neck Pain
Keywords: Biofreeze; Acute Neck Pain; Placebo; chiropractic
MeSH Terms: conditions — Acute Pain; Neck Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The placebo and Biofreeze are in identical containers and only the manufacturer know the contents
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): The experimental group will receive the active product (Biofreeze) over the course of 1 week.
  Interventions: Other: Biofreeze
- Placebo (Sham Comparator): The placebo will use a product created to mimic the topical analgesic Biofreeze over the course of one week. All active ingredients have been removed.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Biofreeze — Biofreeze is a topical analgesic that uses the cooling effect of menthol, a natural pain reliever, to soothe minor muscle and joint pain. The product will be applied 10 minutes prior to manipulation and at home for 4 times a day for 1 week
  Arms: Experimental
Other: Placebo — The placebo is the Biofreeze product with all active ingredients removed. The product will be applied 10 minutes prior to manipulation and at home for 4 times a day for 1 week
  Arms: Placebo

SUMMARY:
The purpose of this study to compare the effect of Biofreeze® versus a Placebo on neck pain, disability, fear avoidance, and range of motion prior to and following cervical manipulation over the course of one week among patients with acute neck pain.

DETAILED DESCRIPTION:
The purpose of this study to compare the effect of Biofreeze® versus a Placebo on neck pain, disability, fear avoidance, and range of motion prior to and following cervical manipulation over the course of one week among patients with acute neck pain. Methods: A convenience sample of 60 acute neck pain patients will be recruited at their initial appointment prior to any therapy being applied. Exclusionary criteria will include pregnancy, cancer, or a corticosteroid injection within the past 2 weeks. Additionally, anyone who has a history of neck surgery will be excluded. Patients will be recruited following their initial examination if they meet the inclusion criteria of pain for less than 2 weeks and be >18 years of age. Eligible patients who agree to participate in the study will complete the informed consent, demographics information questionnaire (including pain medication usage), and paper and pencil instruments that assess their pain, neck disability, and fear avoidance. Cervical range of motion and posture will also be evaluated (T1). After completing the initial paperwork and assessment, patients will then be randomized into either the Placebo [A] (n=30) or Biofreeze® [B] (n=30) group. Both the patient and investigator will be blind to whether topical A or B is the active product. The Biofreeze® group will have Biofreeze® applied directly over the erector spinae muscles of the cervical spine. The Placebo group will have a placebo form of Biofreeze® applied directly over the erector spinae muscles of the cervical spine. After the respective intervention, both groups will wait 10 minutes after the in product is applied to their skin. At the conclusion of the 10 minutes they will again rate their pain (T2). Following the pain rating, all patients will receive a cervical manipulation. Within 5 minutes following the cervical manipulation, all patients will rate their level of pain (T3). Following completion of this rating of pain within 5 minutes following manipulation all subjects will be given the same at-home pain management program. This pain management program will involve applying either Biofreeze® or Placebo to their neck four times per day for the next week based on previous randomization schedule prior to cervical manipulation. All subjects will be instructed to apply the gel they have been assigned directly on top of the erector spinae and site of pain of neck, from inferior to superior to inferior. At one week (T4) patients will complete the paper and pencil instruments and cervical range of motion from the first visit. In addition, at home pain management compliance and pain medication will be documented on a daily basis for the entire week.

ELIGIBILITY:
Inclusion Criteria:

* neck pain for less than 2 weeks and >18 years of age

Exclusion Criteria:

* pregnancy, cancer, or a corticosteroid injection within the past 2 weeks. Additionally, anyone who has a history of neck surgery will be excluded

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Change in Numeric Pain Rating Scale (NPRS) at 1 week | Baseline (T1), 10 minutes after application (T2), immediately following manipulation [15 minutes after application] (T3), 1 week (T4)
Change in Neck Disability Index (NDI) at 1 week | Baseline (T1), 1 week (T4)
Change Cervical Range of Motion at 1 week | Baseline (T1), 1 week (T4)
  Using FDA cleared DorsaVi sensor system to measure cervical flexion, extension, side bending, and rotation

CONTACTS AND LOCATIONS:
Locations (1):
- Sport and Spine Rehab, Landover, Maryland, United States

IPD SHARING:
Plan to Share IPD: No